CLINICAL TRIAL: NCT03065348
Title: A Multimodal Pre- and Intraoperative Approach for Frail Cystectomy Patients. A Prospective Single-arm Matched Case Feasibility Study
Brief Title: Perioperative Multimodal Care for Cystectomy Frail Patient
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of study participants
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CARE-MAC Study
Record Dates: First submitted 2017-02-17; First posted 2017-02-27 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Frail Elderly Syndrome; Bladder Disease; Nutrition Disorders; Cognitive Symptom
Keywords: prehabilitation; nutrition; hydration; cystectomy and urinary diversion; regional anesthesia; cognition
MeSH Terms: conditions — Urinary Bladder Diseases; Nutrition Disorders; Neurobehavioral Manifestations | interventions — Whey Proteins; Immunonutrition Diet

STUDY DESIGN:
Intervention Model Description: First step: pilot study including 20 patients (intervention ) Second step: inclusion of 11 additional patients. Comparison of the intervention group (n=31) with a historical similar population (control group, n=31)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): 1. Around 2 to 4 weeks before surgery:
     * Fried frailty score
     * CARE score assessment
     * NRS Kondrup assessment
     * Plasma albumin and CRP values
     * Start with daily oral whey protein administration until evening before surgery45
  2. Around 5-7 days before surgery:
     - Start with immunonutrition
  3. Evening before surgery:
     * CARE score assessment
     * NRS Kondrup
     * CERAD cognition test assessment
     * Plasma albumin and CRP values, urine specific gravity
     * Carbohydrate loading
     * If urine specific gravity is >1.020 then additional tap water drinking will be encouraged
  4. Day of surgery:
     * Carbohydrate loading
     * Start anesthesia with spinal anesthesia (continuous)
  5. POD 7:
     * CARE assessment
     * CERAD assessment
     * Plasma albumin and CRP values
  6. POD14:
     * CARE assessment
     * Plasma albumin and CRP value
  7. POD 30:
     * CARE assessment
     * NRS Kondrup
     * CERAD assessment
     * Plasma albumin and CRP values
  8. POD 90:
     * CARE assessment
     * NRS Kondrup
     * CERAD assessment
  Interventions: Dietary Supplement: oral whey protein; Dietary Supplement: Immunonutrition; Dietary Supplement: Carbohydrate Drink; Other: Preoperative hydration; Other: continous spinal anesthesia

INTERVENTIONS:
Dietary Supplement: oral whey protein — This substance is specifically formulated to target the nutritional needs of the elderly when they require increased energy and strength, such as following a fall or fracture or for the management of under nutrition and frailty. It provides 300 kcal, 20g of protein and increased levels of vitamin D, calcium. Available in vanilla, caramel and strawberry-biscuit
  Other Names: Resource Whey Protein, Nestlé Health Schweiz
Dietary Supplement: Immunonutrition — This substance is a clinically proven nutritional solution for the dietary management of major elective surgery patients, to improve clinical outcomes, and reduce postoperative complications and length of hospital stay. IMPACT formulation contains omega-3 fatty acids, arginine and nucleotides, and is suitable for use as a sole source of nutrition. Oral IMPACT is a powdered sip feed that provides 303kcal per portion when reconstituted with water (74g powder plus 250ml water) and is enriched with omega-3 fatty acids, arginine, nucleotide, 3 gr of soluble fibre 321mg sodium, 402 mg potassium, 216 mg phosphate per portion.
  Other Names: Oral Impact, Nestlé Health Schweiz
Dietary Supplement: Carbohydrate Drink — Resource® preload™ contains the following elements:
  Per portion à 50gr 47.5 gr carbohydrate, < 10mg sodium, 190kcal
  Other Names: Resource Preload Nestlé Health Schweiz
Other: Preoperative hydration — If urine specific gravity is >1.020 then additional tap water drinking will be encouraged (1% of ideal body weight)
Other: continous spinal anesthesia — Surgery will be performed under continuous spinal anesthesia without general anesthesia

SUMMARY:
Major surgery in the elderly and frail patient is a challenge. Optimal perioperative management is essential for outcome and survival. There is a need for improved multidisciplinary approach to improve postoperative outcome in this patient population at high risk for postoperative morbidity and mortality. Here the investigators will evaluate the implementation of a multimodal prehabilitation program including optimization of nutrition (protein and carbohydrate loading), optimization of preoperative hydration and the use of regional anesthesia during cystectomy and urinary diversion in a series old frail patients and compared/matched them to a historical series of similar patients in terms of early return of quality of life using the Convalescence and Recovery Evaluation (CARE) instrument, cognition, and postoperative morbidity.

The importance of patient-reported health status is well recognized and is a facet of healthcare quality. In addition it is a valuable means for quantitatively measuring the implication of technology adoption for the patient, who typically judges the efficacy of a surgical procedure by whether it improves quality of life.

The objective of this study is to evaluate the implementation of a multimodal prehabilitation program in a series old frail patients and compared them to a historical series of similar frail patients in terms of early return of quality of life, cognition, and postoperative morbidity. The importance of patient-reported health status is well recognized and is a facet of healthcare quality. In addition it is a valuable means for quantitatively measuring the implication of technology adoption for the patient, who typically judges the efficacy of a surgical procedure by whether it improves quality of life.

DETAILED DESCRIPTION:
In industrialized countries the average life expectancy has continuously increased during the last decades and this trend is expected to continue. In Switzerland, a sexagenarian now has a 50% chance, if male, and 70% if female of reaching the age of 80. By 2050, the population of over 80 year-olds will have multiplied 2.7 times in Switzerland. Age is considered the greatest single risk factor for developing cancer, bladder cancer is no exception and typically affects old patients with a median age at the time of diagnosis of around 70. In the US 32% of patients diagnosed with bladder cancer are between 75 and 84. In addition, the prevalence of comorbidities in this old population is very high as hypertension is present in 50-60%, coronary artery disease in 15%, cardiac failure in 15%, dementia in 30%, diabetes in 10-20%, hearing and vision loss in 20-30%. The presence of advanced age, several comorbidities, new acute medical condition (i.e. fracture or newly diagnosed cancer) define the clinical condition of frailty. This medical condition is a consequence of age-related decline in many physiological systems, with defects accumulating with the passage of time (age) resulting in an increased risk of death (ageing).

So surgery and the perioperative period can be exceptionally challenging in old and frail patients due to the presence of comorbidities and age-related physiological changes. In these patients treatment goals should focus on maintaining a good quality of life for the remaining time span by aiming for excellent functional results and if possible long term remission. The gold standard of care today for muscle invasive bladder cancer is pelvic lymph node dissection, cystectomy and urinary diversion which is associated with a high postoperative complication rate (50%). This is probably why today younger age, high stage or grade disease and lower comorbidity are associated with higher odds of receiving radical cystectomy. However, elderly alone should not preclude the indication for radical cystectomy and urinary diversion. In addition there is evidence that the type of anesthesia may impact cognition in old patients. Major cardiac and non-cardiac surgical procedures are known to affect cognitive function. The incidence of postoperative cognitive dysfunction (POCD) varies greatly (4% to 41% after major surgery). POCD may persist being a risk factor for long-term cognitive deterioration.

There is evidence that a multimodal prehabilitation program including optimization of nutrition and mobilisation can improve functional recovery after surgery, resulting in less complications and short length of stay. Optimizing the nutritional status of the frail patients before cystectomy and avoiding general anesthesia could be an alternative to conventional pre- and intraoperative approaches to improve outcome and quality of life, including pain early return of gastrointestinal function cognition and functional activities.

The objective of this study is to evaluate the implementation of a multimodal prehabilitation program including optimization of nutrition (protein and carbohydrate) and hydration combined with the use of regional anesthesia (spinal-epidural anesthesia) during cystectomy in a series old frail patients and compared/matched them to a historical series of similar frail patients in terms of early return of quality of life using the Convalescence and Recovery Evaluation (CARE) instrument, cognition (CERAD test), and postoperative morbidity. As there is a need for a shift in the emphasis towards more patient and recovery-centric measures such as quality of life, the investigators decide to assess the early return of quality of life using the CARE instrument as the primary endpoint. The CARE instrument is a robust multi-dimensional measure of convalescence after major abdominal and pelvic surgery. It has been specifically designed and validated for patients undergoing abdominal and pelvic surgery (like cystectomy) with a high test retest reliability. The CARE instrument covers 4 domains (pain, gastrointestinal, cognition and activity). The importance of patient-reported health status is well recognized and is a facet of healthcare quality. In addition it is a valuable means for quantitatively measuring the implication of technology adoption for the patient, who typically judges the efficacy of a surgical procedure by whether it improves quality of life. The Consortium of Establish a Registry for Alzheimer's Disease (CERAD) test is a widely validated test packet for evaluation of old patients with dementia. However this CERAD test has also been validated in the perioperative setting. It consists of a test battery, including verbal fluency, Boston naming test, word list learning, constructional praxis, word list recall, word list recognition, and mini mental state examination, which can detect subtle changes in cognition. It is easy applicable and the investigators have expertise using this test in a similar cystectomy population.

The investigators will, in a first step, start with a pilot study including 20 patients in order to assess the feasibility of the multimodal approach in the urologic clinic and this population. The sample size for the feasibility endpoint is based on convenience and no a priori calculation was conducted. This number of patients is comparable to published case series illustrating the feasibility of this anesthetic technique for cystectomy patients.

Secondly, the investigators will add 11 patients in the intervention group and then compare this series with a historical series of 31 similar frail and old cystectomy patients. This is based on the CARE results of the historical series (mean CARE score on POD 7 of 50.68 with a SD ± 6.43 and considering a difference of 7 points as clinically relevant with an effect size of 0.7).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* ≥ 75 years old
* Fried frailty score ≥2
* Cystectomy with urinary diversion
* No contra-indication for spinal or epidural anesthesia

Exclusion Criteria:

* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* Women who are pregnant or breast feeding (not applicable as recruitment concerns patients with ≥75 yrs of age)
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* Specific exclusions for the disease under study,
* Specific concomitant therapy washout requirements prior to and/or during study participation,
* Dietary restrictions: milk allergy
* Refusal to regional anesthesia
* Risk of aspiration
* Oral fluid restriction due to any reasons (severe renal insufficiency i.e. GFR < 20ml/min)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change in CARE score | baseline before surgery to postoperative day (POD) 7
  The CARE score is a robust multi-dimensional measure of convalescence after major abdominal and pelvic surgery. The CARE instrument covers 4 domains (pain, gastrointestinal, cognition and activity). The CARE score has been specifically designed and validated for patients undergoing abdominal and pelvic surgery (like cystectomy) with a high test retest reliability ranging from 0.78 to >0.88. The importance of patient-reported health status is well recognized and is a facet of healthcare quality. In addition it is a valuable means for quantitatively measuring the implication of medical treatment for the patient, who typically judges the efficacy of a surgical procedure by whether it improves quality of life

SECONDARY OUTCOMES:
Change in CARE score | from POD 7 to 14, 30 and 90
  see above
Changes in cognition | from baseline (before surgery) to Day 7 and Day 90
  CERAD test performance:
  The Consortium of Establish a Registry for Alzheimer's Disease (CERAD) test is a widely validated test packet for evaluation of old patients with dementia. However this CERAD test has also been validated in the perioperative setting. It consists of a test battery, including verbal fluency, Boston naming test, word list learning, constructional praxis, word list recall, word list recognition, and mini mental state examination, which can detect subtle changes in cognition. It is easy applicable and the investigators have expertise using this test in a similar cystectomy population.
Postoperative complication rate according to Clavien Dindo | within the first 90 day after surgery
  Clavien Dindo complications:
  This is the most widely used classification system for postoperative complications, and is well established in cystectomy patients. An additional more sensitive index has been recently been introduced called Complication Comprehensive Index (CCI) to measure surgical morbidity .
Comprehensive complication index (CCI) | within the first 90 day after surgery
  An additional more sensitive index has been recently been introduced called Complication Comprehensive Index (CCI) to measure surgical morbidity .

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wuethrich, MD, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (1):
- University Hospital Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No